CLINICAL TRIAL: NCT06310070
Title: 3D Printed Personalized Ostomy Appliance
Acronym: 3DPPOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-23-1965
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: 3D Printing; Ostomy; Leakage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Receiving 3D Personalized Ostomy Appliance (Experimental): The personalized ostomy appliances are designed based off of a 3D scan. We will scan your ostomy to create a 3D picture in the computer system that is an exact copy of your ostomy using plastic. We then apply computer aided design (CAD) tools to modify your normal ostomy baseplates.
  Interventions: Device: 3D Printed Personalized Ostomy Appliance

INTERVENTIONS:
Device: 3D Printed Personalized Ostomy Appliance — Study procedures will include getting your stoma scanned, receiving personalized ostomy appliances in the mail, receiving a personalized ostomy template, which will be printed using a 3D printer, in the mail, and completing a daily symptom diary along with a weekly survey for 4 weeks.3D printing is done using a machine that takes the 3D image from the computer and prints a replica of the image using plastic or other materials.

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of using a 3D scan for a personal ostomy appliance. The main question it aims to answer is:

• Whether or not a 3D scan of a stoma reduces leakages and improves patient quality of life in regard to using a personalized ostomy appliance.

Participants will

* Spend 2 weeks with their standard of care ostomy appliance
* Spend 2 weeks with their personalized ostomy appliance made from a 3D scan
* Participate in daily surveys and weekly quality of life surveys conducted over the phone

DETAILED DESCRIPTION:
Formation of an ostomy is an operation that connects a hollow viscus, such as the bowel, to the skin. An ostomy appliance is worn to collect waste around the stoma, the externalized viscus organ. Ostomy appliances are emptied several times a day and are exchanged as infrequently as once per week or as frequently as multiple times per day. Unfortunately, half of all patients with an ostomy will suffer from complications such as peristomal skin breakdown, skin irritation, leaks, and bleeding. Stoma measuring guides are used to measure the ostomy appliance to achieve a well-fit skin barrier and prevent peristomal skin complications. Leaks both dramatically decrease patients' quality of life and result in skin irritation and other complications including infections.

Investigators propose utilizing advances in 3D scanning, computer-aided design (CAD) modeling, and 3D manufacturing to create a personalized ostomy appliance.

Site investigators will develop a 3D personalized ostomy appliance protocol featuring three phases: first, the patient's stoma is scanned using a 3D scanner in CRSudio2; second, the raw scan is edited using personalized variables to create a filtered mesh; third, the filtered mesh is printed to provide an ostomy template to the patient and currently available ostomy appliances are modified using a laser cutter to provide a personalized ostomy appliance to the patient. The selection of commercially available ostomy appliance will be done in coordination with the ostomy nursing team. Based upon the patient's body habitus and stoma, the ostomy nurse will select the recommended appliance that is available at Carilion Clinic. This will be the appliance that is customized using the laser cutter.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* Must have had current ostomy appliance for > 6 weeks - if patients with stomas less than 6 weeks are included, their personalized templates will not be useful once the stoma size has changed after their initial scan.
* Must have experienced > 1 leakage in the week leading up to day of consent. - If patients are not experiencing leakages, then there will be no baseline data to compare effectiveness of the post-3D appliance intervention.
* Participants must be able to consent for themselves
* Access to phone AND computer with internet access. Patient must be able to provide electronic mailing address for e-consent documentation and REDCap surveys.

Exclusion Criteria:

* Concern for patient being able to be reached over the phone or reliable internet access for REDCap survey completion
* Existing peri-stomal skin breakdown including ulceration or mucocutaneous separation.
* Diagnosis of infection around the peristomal region. (erythema is NOT an exclusion criteria)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Leaks | 28 days
  Number of leaks experienced on a daily basis by participant

SECONDARY OUTCOMES:
Number of appliances | 28 days
  Number of ostomy bag changes completed by participant
Overall patient satisfaction | 28 days
  Ostomy Leak Appliance Tool Survey will ask participants to answer questions related to their experiences of leaking within the previous 7 days, including information on the frequency of leakage and emotional impact of how a leak or risk of leakage affected how the participant felt. Participants will answer how they felt, whether they were able to complete usual day to day activities and how they coped by answering on a scale of "All of the time," "Often," "Sometimes," or "Rarely or never."

CONTACTS AND LOCATIONS:
Overall Officials: Farrell Adkins, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States